CLINICAL TRIAL: NCT02335723
Title: Abdominal Septic Shock - Endotoxin Adsorption Treatment (ASSET) - a Double-Blind, Randomized Placebo-Controlled Clinical Investigation With Alteco® LPS Adsorber
Brief Title: ASSET - a Double-Blind, Randomized Placebo-Controlled Clinical Investigation With Alteco® LPS Adsorber
Acronym: ASSET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem to find eligible patients to include
Sponsor: Alteco Medical AB (Industry)
Collaborators: TFS Trial Form Support (Industry); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-CI-01
Record Dates: First submitted 2014-11-28; First posted 2015-01-12 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alteco LPS Adsorber (Active Comparator): Hemoperfusion and Standard therapy
  Interventions: Device: Alteco LPS Adsorber
- Placebo (Placebo Comparator): Placebo and Standard therapy. The placebo comparator device differs from Alteco® LPS Adsorber only in that no peptide component (i.e. active component) has been attached to the matrix.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Alteco LPS Adsorber — Alteco® LPS Adsorber is a Class IIa medical device developed in accordance with existing international standards. Alteco® LPS Adsorber does not contain any pharmaceutical or toxic components.
  Alteco® LPS Adsorber is used for the adsorption of LPS as endotoxins. The capturing component is a specially designed synthetic peptide developed for adsorption of endotoxin. The capturing component has high affinity to Lipid A, i.e. a constant component in the endotoxin molecule, which ensures efficient reduction of endotoxins from different bacterial species.
  Arms: Alteco LPS Adsorber
Device: Placebo — Exactly the same as Alteco LPS Adsorber but no peptide component has been attached to the matrix (i.e. there is no adsorber functionality)
  Arms: Placebo

SUMMARY:
The primary objective of this clinical investigation is to investigate the feasibility and possible benefits of the Alteco® LPS Adsorber in treating patients with septic shock with presumed endotoxemia of abdominal or urogenital origin.

DETAILED DESCRIPTION:
OVERALL CLINICAL INVESTIGATION DESIGN:

This is a multicentre, stratified, parallel, double-blinded, randomized, feasibility clinical investigation of the Alteco® LPS Adsorber.

Subjects will be enrolled in an adaptive fashion with up to two interim analyses, and the possibility of recruiting additional patients, in order to establish an indication of the feasibility of treating a target population of subjects with septic shock and endotoxemia.

Subjects will be stratified in accordance with the origin of their infection, i.e. abdominal or urogenital sepsis. Subjects in each stratum will receive either:

* LPS Adsorber group (i.e. investigational medical device [IMD] group): current best practice in combination with Alteco® LPS Adsorber treatment, OR
* Placebo device group (i.e. comparator group): current best practice in combination with placebo adsorber treatment.

Allocation to either treatment arm will be performed in a 1:1 ratio. Upon enrolment (i.e. pre-treatment phase), subjects admitted to the ICU with suspected endotoxemia will be screened for fulfilment of the "Illness Severity Criteria" confirming early stage severe sepsis.

Within six (6) hours of enrolment, subjects who also fulfil the "Treatment Criteria" confirming septic shock will be eligible for randomization.

Randomization to either of the treatment groups will be performed as close as possible to start of treatment with the Alteco® LPS Adsorber or placebo device.

Treatment with LPS Adsorber or placebo device must be initiated within six (6) hours (Day 1) following fulfilment of the "Treatment Criteria". A second device treatment will be performed 24 hours after the end of the first device treatment on Day 2, as long there is no evidence that treatment with the investigational device will not be beneficial or will indicate an unnecessary risk for subjects (for example, the subject is vasopressor support-free).

Initially: 20 abdominal sepsis subjects (Stratum A) and 12 urogenital sepsis subjects (Stratum B) Optional: additional 12 subjects (abdominal, urogenital or both) after interim analysis decision.

ELIGIBILITY:
Inclusion Criteria:

Illness severity criteria: At enrolment subjects must meet inclusion criteria #1 through #3 listed below to be eligible to enter the clinical investigation:

1. Subjects must have suspected severe infection of abdominal or urogenital origin for which the subject is receiving intravenous antimicrobial therapy as the main reason for organ support
2. Subjects, males or females, must be 18 years or older.
3. Subjects or legally acceptable representatives, as appropriate, are willing and able to provide signed informed consent.

   Treatment criteria: Prior to randomization, subjects must meet all inclusion criteria (#4 through #7) listed below to be assigned to a treatment group:
4. Appropriate vascular access must have been obtained.
5. Subjects must have received ≥ 30 mL/kg of intravenous fluid within the six (6) hours prior to randomization.
6. Subjects must have plasma/serum lactate >2 mmol/L despite adequate resuscitation AND a continuous requirement for vasopressor support
7. Subjects must be able to initiate the clinical investigation intervention within 12 hours of fulfilment of the illness severity criteria.

Exclusion Criteria:

1. Subjects who meet any of the exclusion criteria listed below will NOT be permitted to enter the clinical investigation: Sepsis-induced organ dysfunction for longer than 12 hours prior to the time-point for achieving "Illness severity criteria fulfilled"
2. Vasopressor therapy (at any dose) for longer than 12 hours (not included the time spent in the operation theatre) prior to the start of treatment with the investigational device.
3. Pre-existing uncorrectable medical condition as:

   * Poorly controlled neoplasms or hematologic disease (i.e. indication of disseminated cancer outside the suspected primary tumour and hematologic disease not in remission,
   * End-stage cardiac disease,
   * Cardiac arrest requiring cardiopulmonary resuscitation or with pulseless electrical activity or asystole within the past 7 days
   * End-stage lung disease
   * End-stage liver disease
   * HIV/AIDS with known end-stage processes
   * Other uncorrectable medical condition(s) deemed by the Clinical Investigator to hinder the subject to adhere to the fulfilment of the activities described in the Clinical Investigation Plan.
4. Extreme illness, i.e. subjects is moribund and death is perceived to be imminent (within 24 hours).
5. Recent or current participation (≤ 30 days) in another interventional sepsis trial.
6. Recent or current treatment (≤ 30 days) with an adsorption product, including Alteco® LPS Adsorber.
7. Treatment with an investigational medicinal product for any indication within the last 30 days before enrolment in the clinical investigation.
8. Pregnancy.
9. Contraindications to the use heparin or protamine
10. Other abdominal inflammatory conditions
11. Perforation of hollow organ linked to trauma within 48 hours before enrolment in the clinical investigation.
12. Laparotomy reveals isolated gastric ulcer.
13. Subjects and/or their immediate family are directly affiliated to investigative site personnel in this clinical investigation. (Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Characterization of all reported USADEs and ASADEs. | 6-28 days

SECONDARY OUTCOMES:
Relative change from baseline in plasma endotoxin (p-endotoxin) levels during (i.e. at 2 hours) and immediately after end (i.e. at 6 hours) of treatment with device, on both Day 1 and Day 2. | 2 days
Relative change from baseline in SOFA score | 6-28 days
Relative change from baseline in renal function | 6-28 days
  Renal function is assessed by: S-creatinine, P-Cystatin C, P-Urea, eGFR, KDIGO stage, Fluid balance, and Daily urinary output
Relative change from baseline in liver function | 6-28 days
  Liver function is assessed by: Prothrombin complex INR, P-Albumin, and P-Bilirubin
Relative change from baseline in circulatory support | 6-28 days
  Circulatory support is assessed by: Vasopressor load, Inotropic score, MAP, Vasopressor dependence index, P-Lactate, Blood gas, and Vasopressor-free days.
Relative change from baseline in respiratory support | 6-28 days
  Respiratory support is assessed by: PaO2, FiO2 and PaO2/FiO2 ratio, Positive and expiratory pressure, Peak pressure, Tidal volume and minute volume, Respiratory rate, Pa CO2, Respiratory support need as measured by means of ventilator-free days until day for ICU discharge
Relative change from baseline in ICU mortality | 6-28 days
Relative change from baseline in ICU length of stay | 6-28 days
Clinical outcome during stay at Hospital following ICU-discharge of the total extension of renal support | 6-28 days
Clinical outcome during stay at Hospital following ICU-discharge of 28-day mortality | 6-28 days
Clinical outcome during stay at Hospital following ICU-discharge of hospital length of stay up to 28 days | 6-28 days
Levels of inflammatory response biomarkers | 6-28 days
Determination of the molecular components extracted from blood circulation and captured in Alteco® LPS Adsorber. | 6-28 days
  This is an exploratory outcome, there will be a screening of which molecules that have been captured.
Characterization of all reported AEs (regardless of attribution), ADEs, and device deficiencies | 6-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rubertsson, Professor, Principal Investigator — Uppsala University Hospital
Locations (6):
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus, Oslo
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipcsey M, Tenhunen J, Pischke SE, Kuitunen A, Flaatten H, De Geer L, Sjolin J, Frithiof R, Chew MS, Bendel S, Kawati R, Larsson A, Mollnes TE, Tonnessen TI, Rubertsson S. Endotoxin Removal in Septic Shock with the Alteco LPS Adsorber Was Safe But Showed no Benefit Compared to Placebo in the Double-Blind Randomized Controlled Trial-the Asset Study. Shock. 2020 Aug;54(2):224-231. doi: 10.1097/SHK.0000000000001503. PMID 31880758
- [Derived] Lipcsey M, Tenhunen J, Sjolin J, Frithiof R, Bendel S, Flaatten H, Kawati R, Kuitunen A, Tonnessen TI, Rubertsson S. Abdominal Septic Shock - Endotoxin Adsorption Treatment (ASSET) - endotoxin removal in abdominal and urogenital septic shock with the Alteco(R) LPS Adsorber: study protocol for a double-blinded, randomized placebo-controlled trial. Trials. 2016 Dec 8;17(1):587. doi: 10.1186/s13063-016-1723-4. PMID 27931259